CLINICAL TRIAL: NCT05236179
Title: Patient Survey on Integrative Therapy Methods - a Cross-sectional Study of Hospital Inpatients
Brief Title: Survey of Inpatients on Integrative Therapy Methods
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PAT_01
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Patient Satisfaction and Experience With Integrative Therapies
Keywords: Integrative therapies; Anthroposophic medicine; Overall patient satisfaction; Inpatients; Survey
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Integrative therapies — Integrative therapy methods used at the Filderklinik, such as music therapy, therapeutic painting, therapeutic sculptural forming, speech therapy, eurythmy therapy, rhythmical massage, external applications, coloured light therapy

SUMMARY:
Observational study of general patient satisfaction and inpatients' experiences with integrative therapies. The study recruits inpatients of the Filderklinik, an anthroposophic hospital in southwestern Germany. The aim is to assess overall patient satisfaction and inpatients' experiences with integrative therapies at the Filderklinik.

DETAILED DESCRIPTION:
This is a cross-sectional study to investigate general patient satisfaction and inpatients' experiences with integrative therapies in an anthroposophic hospital. Participants will be recruited at the Filderklinik, a hospital in southwestern Germany that uses anthroposophic medicine (AM) on a broad basis. Inpatients who have received at least 10 treatments with one or more of the different integrative therapy methods will be asked for their willingness to participate. After providing written informed consent, participants will complete a questionnaire on integrative therapies received and overall patient satisfaction. In addition, data from the clinic database will be analyzed and cross-checked with the questionnaire data to verify and specify information about the participating sample. The focus of the study is to assess general patient satisfaction and experience with integrative therapy methods among inpatients at the Filderklinik.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Filderklinik inpatient who had at least 10 treatments with one ore more of the integrative therapy methods
* Age 18 years or older

Exclusion Criteria:

* Insufficient German language skills
* Legally incapacitated patients
* Patients who are physically incapable of giving written consent
* Patients in isolation wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients of the Filderklinik who have received at least 10 treatments with one or more of the various integrative therapy methods used at the Filderklinik.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction, ZUF-8 total score | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient satisfaction, measured with the ZUF-8 patient satisfaction questionnaire, a validated questionnaire (German language) with 8 items related to overall patient satisfaction associated with an inpatient hospital stay. Items are rated on 4-point scales from positive to negative (no "neutral" position), with 1 being the least positive and 4 being the most positive value (total scale range 8-32). In the current study, the ZUF-8 is part of the comprehensive "Special Therapy Procedures" questionnaire, which covers all outcome measures not retrieved from the clinic database.

SECONDARY OUTCOMES:
Diagnoses | Assessing the entire duration of the hospital stay, an average of 7 days.
  Diagnoses of each patient documented in the clinic database.
Therapies | Assessing the entire duration of the hospital stay, an average of 7 days.
  Therapies that were prescribed to each patient, as documented in the clinic database.
OPS codings | Assessing the entire duration of the hospital stay, an average of 7 days.
  OPS codings for each patient documented in the clinic database. OPS = Operationen- und Prozedurenschlüssel, German modification of the ICPM (International Classification of Procedures in Medicine).
Inpatient admitting department | At the time of admission to the Filderklinik, at the beginning of hospitalization (an average of 7 days).
  Department of the Filderklinik to which the patient was admitted for the inpatient stay.
Integrative therapies according to clinic database | Assessing the entire duration of the hospital stay, an average of 7 days.
  Integrative therapies that were prescribed to each patient, as documented in the clinic database.
Patient experience with music therapy | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the music therapy prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with therapeutic painting | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the therapeutic painting prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with therapeutic sculptural forming | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the therapeutic sculptural forming prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with speech therapy | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the speech therapy prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with eurythmy therapy | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the eurythmy therapy prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with rhythmical massage | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the rhythmical massage prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with external applications | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the external applications prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with coloured light therapy | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the coloured light therapy prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with the timing of integrative therapies | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with the timing of the integrative therapies prescribed to them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Patient experience with therapy plan communication | Assessing the entire duration of the hospital stay, an average of 7 days.
  Patient experience with communication about the therapy plan that was set up for them, assessed with the "Special Therapy Procedures" questionnaire. The questionnaire records general patient satisfaction and patient experience with the integrative therapy methods at the Filderklinik and asks for aspects of organization and procedure as well as the therapy itself. Answers are given on a 5-point Likert scale ranging from "I fully agree" to "I fully disagree", with "I fully agree" representing positive ratings.
Difference in patient satisfaction: prior experience with AM vs. no prior experience with AM | Assessing the entire duration of the hospital stay, an average of 7 days.
  Difference in patient satisfaction between the group of patients who had prior experience with AM and the group who had no prior experience with AM, measured with the ZUF-8 questionnaire. ZUF = "Zufriedenheit" = satisfaction. ZUF-8 = patient satisfaction questionnaire, a validated questionnaire (German language) with 8 items related to overall patient satisfaction associated with an inpatient hospital stay. Items are rated on 4-point scales from positive to negative (no "neutral" position), with 1 being the least positive and 4 being the most positive value (total scale range 8-32).
Difference in patient satisfaction: Filderklinik chosen for treatment with AM vs. Filderklinik chosen for other reasons | Assessing the entire duration of the hospital stay, an average of 7 days.
  Difference in patient satisfaction between the group of patients who chose the Filderklinik because they request treatment with AM and the group who chose the Filderklinik for other reasons, measured with the ZUF-8 questionnaire. ZUF = "Zufriedenheit" = satisfaction. ZUF-8 = patient satisfaction questionnaire, a validated questionnaire (German language) with 8 items related to overall patient satisfaction associated with an inpatient hospital stay. Items are rated on 4-point scales from positive to negative (no "neutral" position), with 1 being the least positive and 4 being the most positive value (total scale range 8-32).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr, Study Director — ARCIM Institute Academic Research in Complementary and Integrative Medicine
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.